CLINICAL TRIAL: NCT05017909
Title: The Effect of Education Given to Primipara Pregnancy With Two Different Methods (Face-To-Face/ Web-Based) in the Last Trimester on Their Acquisition of the Mothering Role
Brief Title: The Effect of Different Education Techniques on the Acquisition of the Mothering Role
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Imren ARPACI, PHD Student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IARPACI
Record Dates: First submitted 2021-05-24; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Gaining the Role of Motherhood in Primipara Pregnancy (Focus)
Keywords: Primipara Pregnancy; Role of Motherhood; Web-Based Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): 3-week web-based education group
  Interventions: Behavioral: Web based education
- Experimental Group 2 (Experimental): 3-week face to face education group
  Interventions: Behavioral: Face to face education
- Control Group (Active Comparator): Uneducated group
  Interventions: Behavioral: No education

INTERVENTIONS:
Behavioral: Face to face education — Face to face education techniques on the acquisition of the mothering Role
  Arms: Experimental Group 2
Behavioral: Web based education — web based education techniques on the acquisition of the mothering Role
  Arms: Experimental Group 1
Behavioral: No education — Control group will not be educated
  Arms: Control Group

SUMMARY:
The research consists of two stages.

First Stage: It is the development of the scale for gaining the role of motherhood in primiparas according to the scale development stages. In order to define the subject and determine the scope, the content analysis will be determined by interviewing the sample group that will not be included in the pilot application and the final scale application and the primipara people with similar characteristics. As a result, the item pool will form the basis together with the literature. An item pool related to gaining the role of motherhood will be created, the opinions of experts will be taken to evaluate the scope and appearance validity of the scale, and adjustments will be made in the item pool according to expert opinions.

In order to determine the validity and reliability of the scale, half of the participants will be tested-retested. The internal consistency reliability of the scale will be determined by the Cronbach Alpha reliability coefficient. In addition, Edinburgh Postpartum Depression Scale (EDDS) and Mother-Infant Attachment Scale (MIAS), which are similar scales, will be used in the scale development phase for the validity of the scale.

Second stage: The training consisting of 3 modules is planned. MODULE: Mother Module MODULE: Infant Module MODULE: Breastfeeding Module

At this stage of the study, pregnant women who meet the sampling criteria will be divided into groups. The determination of the groups will be according to the Randomized numbers table. Pregnant women who will enter the web-based training group (Experimental group 1), Face-to-face training group (Experimental group 2) and the control group will be determined.

The personal information form containing the socio-demographic data and the final scale developed to gain the role of motherhood in primiparas will be applied to the participants who volunteered to participate in the study.

Experimental Initiative: A web-based and face-to-face training program will be planned and implemented as separate groups for the sampled participants.

Post-Test Application of the Final Scale: The final scale, which was developed to gain the role of motherhood in primiparas, will be administered to the participants in the sample group as a post-test on the 40th day.

By analyzing the data obtained, the effectiveness of the scale and the difference between the pre-test scores of the participant group after the training program will be examined.

DETAILED DESCRIPTION:
The research was planned methodologically and experimentally. A motherhood role acquisition scale will be developed as a methodological study, and web-based and face-to-face training will be given experimentally. The effect of the training given on the acquisition of the role of mother will be determined.

The research will be conducted between September 2021 and September 2022.

The Universe and Sample of the Research; the population of the research will be all primiparous pregnant women who meet the criteria for participation in the study and volunteer to participate in the study in two different Family Health Centers (FHC) affiliated to Gaziantep Provincial Health Directorate and Private Dr. Tuncay Yüce Gynecology and Obstetrics Clinic.

The sample of the first stage of the research; determined by the number of items in the scale. When we examine the literature, it is seen that there will be 5-10 times as many participants as the number of items, and the sample size should be at least 50 in the data for which factor analysis will be applied.

The sample of the second phase of the research; With G-Power, it was determined that there were 42 people in the experimental 1 group, 42 in the experimental 2 group, and 42 in the control group at 80% power, 5% error and 95% confidence interval. Data collection will take place between September 2021 and May 2022.

Location and Characteristics of the Research; The research will be carried out between December 2021 and May 2022 with primiparous pregnant women in two different Family Health Centers (ASM) affiliated to Gaziantep Provincial Health Directorate and Private Dr. Tuncay Yüce Gynecology and Obstetrics Clinic. There are 10 Family Medicine units in total in two centers, and there are baby care rooms and breastfeeding rooms where training can be provided for pregnant women in Family Health Centers.

Application of Research

Under the guidance of the literature, an item pool will be created and the content validity of the scale will be determined by taking the opinions of field experts. Care will be taken to ensure that the sample size is at least 5 times the number of items. After the approval of the ethics committee, the written consent of the primiparous pregnant women who volunteered to participate will be obtained and they will be asked to respond to the data collection tool. The data obtained will be analyzed, and the final form will be created by selecting items with high reliability according to the results obtained.

For the last form, the sample size will be calculated according to the minimum sample size formula to represent the population. The final form will be applied after obtaining written permission from the participants who volunteered to participate in the research. The obtained data will be analyzed and interpreted.

Experimental group 1

The purpose of the study will be explained to the pregnant women in the experimental group 1, and those who accepted to participate in the study and who met the criteria of the study would have to fill in the personal information form prepared by the researcher as a pre-test form, which includes socio-demographic data, and the scale developed to gain the role of motherhood. Afterwards, a 3-week training will be applied on the created web page, and the scale developed to give mothers the role of motherhood as a post-test will be applied in the first 40 days following the birth of expectant mothers.

Experimental group 2

The purpose of the study was explained to the pregnant women in the experimental group 2, and those who accepted to participate in the study and who met the criteria of the study would be asked to fill in the personal information form prepared by the researcher, containing the socio-demographic data as a pre-test form, and the scale developed to gain the role of motherhood in Primiparas. Then, a 3-week face-to-face training will be applied, and the scale developed to give mothers the role of motherhood as a post-test will be applied to mothers in the first 40 days following their birth.

Control group

The purpose of the study will be explained to the pregnant women in the control group, and those who agree to participate in the study and who meet the criteria of the study will be asked to fill in the personal information form containing their socio-demographic data as a pre-test form prepared by the researcher, and the scale developed to gain the role of motherhood in Primiparas. The pregnant women in the control group will not be trained, and the scale developed to give mothers the role of motherhood will be applied as a post-test in the first 40 days following their birth.

Educational subjects

The training consists of 3 modules.

1. MODULE: Mother Module
2. MODULE: Baby Module
3. MODULE: Breastfeeding Module

Data Collection Tools

The data during the scale development phase will be collected using the "Draft Scale for Acquiring the Role of Motherhood" form determined in the item pool, the data collection form developed by the researcher, and the Edinburgh Postpartum Depression Scale (EDDS) and the Mother-Infant Attachment Scale (MIAS). The data in the second stage will be collected using the "Scale for Acquiring the Role of Motherhood " and the data collection form developed by the researcher.

ELIGIBILITY:
Inclusion Criteria

* Having a primiparous pregnancy,
* In the last trimester of pregnancy,
* At least primary school graduate,
* Able to read and understand Turkish,
* Use the internet actively and regularly access the website and receive training,
* Do not have any physical, mental or social problems that may prevent participation in face-to-face or web-based education and pregnant women who accepted the study will be included in the study.

Exclusion Criteria

* Pregnant women who cannot access the website,
* Have any congenital defect in their baby,
* Experience mother-baby separation,
* Want to leave the research before the end of the research will not be included in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The effect of education on the role of motherhood | 1 year and 6 months
  As a result of our research, a motherhood role acquisition scale will be developed. This developed scale will be applied to pregnant women in the last trimester. By providing web-based or face-to-face training, it will be determined which training method has a positive or negative effect on gaining the role of motherhood.

CONTACTS AND LOCATIONS:
Overall Officials: Feride Yiğit, Study Director — Hasan KU

IPD SHARING:
Plan to Share IPD: No